CLINICAL TRIAL: NCT06068335
Title: Innate Immunity in Allergic Asthma
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: CR00001150
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Asthma
Keywords: allergy; Immunity; Healthy; respiratory; ENT
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to determine whether a potential type 2 signature, obtained through stimulation of cell lines with various allergens in vitro, correlates with an allergic or asthmatic disease state ex vivo. This type 2 signature will be multi-hierarchical in nature and will be comprised cell surface receptor expression, pathway activation, and gene upregulation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age
* no history of allergic disease (healthy controls), have clinically diagnosed allergies, or have clinically diagnosed asthma.

Exclusion Criteria:

* Pregnant women and prisoners will be excluded from the study.
* Individuals currently suffering from any acute infections and those known to suffer from light-headedness will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will require 100 participants, with a third ideally falling within each category (healthy, allergic, or asthmatic)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
To determine which parameters of the established type-2 signature obtained in vitro is significantly different between healthy controls, allergic individuals, and asthmatic individuals ex vivo. | 1 year

SECONDARY OUTCOMES:
To determine ex vivo whether any of the identified disease-specific type-2 parameters can be modified (brought back to healthy control levels) through the use of investigational compounds. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Justine T Tigno-Aranjuez, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No